# Effect of Single Dose Intravenous Dexamethasone on Postoperative Pain and Complications in Jaw Surgery Under General Anesthesia

**DATE: JANUARY,1,2024** 

Funda ARUN, MD, PhD, Assis. Professor. Selcuk University Faculty of Dentistry, Department of Pedodontics, Division of Anesthesia, Konya, TURKEY.

Emine TASKIN, Dt., Selcuk University Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Konya, TURKEY. https://orcid.org/0009-0000-4846-622X

Hasan KUCUKKOLBASI, PhD, Professor. Selcuk University Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Konya, TURKEY. https://orcid.org/0000-0002-7769-8537

Corresponding Author

Assis. Prof. Funda ARUN

Selcuk University Faculty of Dentistry

Department of Pedodontics Division of Anesthesia,

Alaaddin Keykubat Campus, 42130

Selcuklu, Konya, Turkey

Tel: 0090 5327494542

Email. funda.arun@selcuk.edu.tr

https://orcid.org/0000-0001-7345-0318

#### Introduction

Common postoperative concerns after maxillofacial surgeries, like large cyst enucleation and impacted tooth extractions, include pain, facial swelling, and restricted mouth opening. These issues stem from the inflammatory response following surgical tissue injury [1]. Successfully managing these challenges is crucial for ensuring patient comfort and recovery, as it directly affects their daily routines [2]. Various interventions (local anesthetics, analgesics, corticosteroids) have been used to minimize these inflammatory responses. Corticosteroids are commonly administered interventions for their powerful anti-inflammatory effects in surgery [1].

Dexamethasone (DXM) is one of the corticosteroid medications that has been used in oral and maxillofacial surgery to relieve the postoperative inflammation associated with surgical trauma. DXM works by blocking inflammatory mediators, decreasing capillary dilation, and modifying the production of prostaglandins and leukotrienes [3]. DXM suppresses neuropeptide release, such as calcitonin gene-related peptide and substance P, from nerve endings after tissue damage injury [4]. These actions make dexamethasone an effective choice for managing postoperative acute inflammatory responses.

Intravenous (IV) administration of DXM has been utilized during surgeries conducted under general anesthesia (GA) [5]. The effects of IV DXM typically appear about 1 to 2 hours after administration, as it takes some time to cross cell membranes and begin influencing gene transcription. With a long biological half-life of 36 to 72 hours, just one dose can help maintain cortisol levels for up to an entire week [6]. DXM is crucial in preventing the body's stress defenses from becoming overly intense, which can greatly support a smoother recovery process [7].

DXM is frequently administered to reduce postoperative complications, including pain and facial swelling, especially in procedures like third molar removals and cyst enucleations. However, the extent of its impact on postoperative outcomes, including pain intensity and secondary complications, requires further investigation. In the literature, cases involving the perioperative use of steroids are either performed under local anesthesia or combined with an analgesic/anti-inflammatory drug [8, 9]. These studies frequently fail to specify the type or dosage of local anesthetic. Since local anesthetics with epinephrine are widely used in dentistry due to their vasoconstrictive properties, their pharmacological effects, including secondary anti-inflammatory outcomes, must be carefully considered. Since local anesthetics with epinephrine are commonly used in dentistry, the secondary anti-inflammatory effect of epinephrine due to its vasoconstrictive properties has been overlooked in previous research [10].

This study aims to evaluate the effect of a single-dose IV DXM on postoperative pain and other complications in compacted tooth and cyst enucleation procedures performed under GA.

This single-center prospective observational study was conducted in Selcuk University Faculty of Dentistry after the permission of the Institutional Ethical Committee (2024,269) and registered at clinicaltrials.gov (). Written informed consent for the study inclusion was obtained from all patients under the Declaration of Helsinki. The study included 90 patients with large cyst enucleation or complex impacted tooth extraction under general anesthesia from June 2024 to December 2024. Participants were aged 18 to 65, had ASA physical status I-II, and underwent split-mouth surgery. Patients undergoing corticosteroid therapy for any reason, as well as those with systemic inflammatory or rheumatological conditions, bilateral cysts, or bilateral impacted teeth that require extraction, were excluded from the study.

Standard intraoperative monitoring was applied, including SpO2, ECG, non-invasive blood pressure, and end-tidal CO2. GA was induced with sodium thiopental (3 mg/kg), rocuronium bromide (0.6 mg/kg), and fentanyl (1.5-2 mcg/kg) and maintained using a mixture of 50% oxygen (O2), 50% air, sevoflurane (2%), and remifentanil (0.05–2 µg/kg/min) infusion. All patients were intubated with appropriately sized endotracheal tubes. Following sterilization and draping, the maxillofacial surgery team applied local Articaine HCl with Epinephrine) to the surgical area and proceeded with the procedure. At the end of the procedure, patients received a single IV dose of DXM (0.1 mg/kg) and pantoprazole (40 mg) before being extubated and transferred to the postoperative recovery unit. Postoperative pain was assessed using the Visual Analog Scale (VAS), with scores categorized as <3: mild pain, 3–6: moderate pain, and >6: severe pain. Patients received an analgesic 50 mg Dexketoprofen IV when the VAS score was >3. All patients were discharged from the hospital on the day of surgery.

Follow-up assessments were conducted on postoperative days 1st, 2nd, and 7th by a blinded clinician not involved in the surgical procedures. Facial swelling was quantified using Daniel Lim's methodology, measuring key facial landmarks pre- and postoperatively and calculating the percentage change. The swelling was classified as Grade 0: <3%, Grade I: 3–6%, Grade II: 6–12%, Grade III: >12%. Mouth opening was evaluated using a dental caliper to measure inter-incisal distance, categorized as Grade 0: >2.5 cm (no trismus), Grade I: 2–2.5 cm (mild trismus), Grade II: 1–2 cm (moderate trismus), Grade III: <1 cm (severe trismus).

#### Statistical Analysis

Data were analyzed using SPSS 20.0. Continuous variables were tested for normality using the Kolmogorov-Smirnov test and reported as mean  $\pm$  SD or median values as appropriate. Categorical variables were presented as frequencies and percentages. Group comparisons were performed using t-tests or Mann-Whitney U tests, with p<0.05 considered statistically significant.

# BİLGİLENDİRİLMİŞ GÖNÜLLÜ OLUR FORMU (Informed Consent Form)

#### ARAŞTIRMANIN ADI (ÇALIŞMANIN AÇIK ADI):

GENEL ANESTEZİ ALTINDA ÇENE CERRAHİSİNDE İNTRAOPERATİF TEK DOZ İNTRAVENÖZ DEKSAMETAZONUN POSTOPERATİF AĞRI VE KOMPLİKASYONLAR ÜZERİNE ETKİSİ

Bu çalışma, bir bilimsel araştırmadır. Çalışmaya, katılmak isteyip istemediğinize karar vermeden önce araştırmanın neden yapıldığını, bilgilerinizin nasıl kullanılacağını, çalışmanın neleri içerdiğini ve olası yararları ile risklerini doğru anlamanız önemlidir. Lütfen aşağıdaki bilgileri dikkatlice okumak için zaman ayırınız.

ÇALIŞMANIN AMACI NEDİR? Bu çalışmada Diş Hekimliği Fakültesi'nde, genel anestezi altında çene kistleri ve gömülü diş çekimleri nedeniyle ameliyat edilen hastalara ameliyat sırasında rutin olarak uygulanan intravenöz (İV) deksametazonun, ameliyat sonrası ağrı ve oluşabilecek diğer komplikasyonlar (yüzde ödem, kısıtlı ağız açıklığı) üzerine etkilerini gözlemlemeyi amaçladık.

# ÇALIŞMADA UYGULANACAK TEDAVİLER/İŞLEMLER NELERDİR? (ÇALIŞMANIN YÖNTEMİ NEDİR?

Çalışmamızda size ameliyatınız ve ameliyat sonrası kontrol muayeneleriniz haricinde bu çalışma kapsamında herhangi bir ek tedavi ya da işlem yapılmayacaktır. Ameliyatınızın yapılabilmesi için size genel anestezi verilecektir. Genel anesteziden uyandıktan sonra ameliyathanemizde bulunan Hasta Derlenme Bölümünde anestezi doktoru ve hemşire gözetiminde tamamen anestezi etkisi geçene kadar izlenip, aynı gün içinde taburculuk işleminiz yapılacaktır. Taburculuk öncesi Ağız, Diş ve Çene Cerrahisi bölümünden ameliyatınızdan sorumlu diş hekimleri kontrol muayenenizi yapacak ve reçetenizi oluşturacaktır. Evde doldurmanız için size bir Evde Ağrı İzlem Formu verilecek ve ertesi gün yapılacak kontrol muayenesine bu formu getirmeniz istenecektir. Ameliyat sonrası ağrı, kullandığınız ilaçlar ve klinik muayene bulgularınızı değerlendirerek ameliyat esnasında rutin olarak uygulanan deksametazon adlı ilacın ağrı, ağız açıklığı ve yüzde oluşabilecek ödeme etkilerini gözlemlemeyi amaçlıyoruz.

#### ÇALIŞMANIN KAPSAMI NEDİR?

Çalışmamız genel anestezi altında maksillada en fazla yarım çene büyüklüğünde (tek taraflı) kist eksizyonu veya gömülü diş çekimi yapılacak olan tüm erişkin hastaları içermektedir. Çalışmamızda deneysel herhangi bir işlem ya da uygulama yapılmayacaktır.

## ÇALIŞMA SÜRESİ NE KADARDIR?

Çalışmamızın 1 yıl içerisinde tamamlanmasını planlıyoruz.

## ÇALIŞMAYA KATILMASI BEKLENEN TAHMİNİ GÖNÜLLÜ SAYISI NEDİR?

Çalışmamıza 60 hasta gönüllünün katılımını bekliyoruz.

ÇALIŞMADA BENİM NE YAPMAM GEREKİYOR? Çalışmaya katılmayı gönüllülük içerisinde kabul ettiğiniz taktırde size taburcu olduğunuzda 'Evde Ağrı İzlem Formu' verilecek, bu formun doğru bir şekilde doldurulup 1. Gün yapılacak kontrol muayenesine getirmeniz istenecektir. Bu süreçte elde edilecek bilgilerinizin değerlendirilmesine izin vermeniz ve bu formu okuyup imzalamanız gerekmektedir.

#### BU ÇALIŞMAYA KATILMAK ZORUNDA MIYIM?:

Çalışmaya katılıp katılmamak tamamen sizin serbest iradenize bırakılmıştır. Eğer çalışmaya katılmaya karar verirseniz imzalanmanız için size bu "Bilgilendirilmiş Gönüllü Olur Formu" verilecektir. Katılmaya karar verirseniz, çalışmadan herhangi bir zamanda ayrılmakta özgürsünüz. Bu durum sizin aldığınız tedavinin standardını etkilemeyecektir, gereken her türlü tedavinize devam edilecektir.

Belirtelim ki, çalışmayı yürüten sorumlu araştırmacı (Çalışma Doktoru) çalışmaya katılımınızın devam etmesinin sizin yararınıza olmadığına karar verebilir ve sizin faydanız için sizi çalışmadan çıkarabilir.

Çalışmadan çıkarılmanız; çalışmaya katılmaya uygunluk kriterlerine artık uymamanız veya herhangi bir şekilde sağlığınızın riske girmesi nedeniyle, doktorunuzun çalışmada yer almanızı durdurmaya karar vermesi durumunda veya araştırıcılar sizinle artık temasa geçemediği durumlarda söz konusu olacaktır.

# ÇALIŞMAYA KATILMA İLE BEKLENEN OLASI YAN ETKİLER VE RİSKLER NELERDİR?

Çalışmaya katılmanız durumunda, katılmaktan kaynaklanabilecek herhangi bir yan etki veya risk durumu bulunmamaktadır.

#### CALISMAYA KATILMANIN OLASI YARARLARI NELERDİR?

Çalışmaya katılmanız durumunda kişisel bir yarar elde etmeyeceksiniz.

### ÇALIŞMAYA KATILMANIN MALİYETİ NEDİR?

Bilimsel çalışmaların maddi kaygılarla yürütülmemesi ilkesi gereğince, bu çalışmaya katılmak için bir ödeme yapmanız gerekmez. Katılımınız karşılığında size de bir ödeme yapılmayacaktır.

#### KİŞİSEL BİLGİLERİM NASIL KULLANILACAK?

Bu formu imzalayarak araştırma doktorunuzun ve onun kadrosunun çalışma için sizin kişisel bilgilerinizi (Çalışma Verileri) toplamalarına ve kullanmalarına onay vermiş olacaksınız. Doğum tarihiniz, cinsiyetiniz gibi tüm kişisel çalışma verilerinizin kullanımı ile ilgili verdiğiniz bu onay kural olarak süresiz geçerli olup bunun herhangi bir sona erme süresi yoktur. Eğer verilerinizin kullanılmamasını istiyorsanız doktorunuzu haberdar ederek bu onayınızdan her zaman vazgeçebilirsiniz.

Çalışma yapan araştırmacılar, etik kurul ve ilgili sağlık otoriteleri gerektiğinde sizin tıbbi kayıtlarınıza doğrudan ulaşabilecektir, fakat bu bilgiler gizli tutulacak kamuoyu ile paylaşılmayacaktır. Çalışmanın sonuçları tıbbi yayınlarda yayınlanabilir, ancak sizin kimlik bilgileriniz bu yayınlarda gizli tutulmaya devam edecektir.

Doktorunuzdan, toplanan çalışma verileriniz hakkında her zaman bilgi isteme hakkına sahipsiniz. Aynı zamanda bu verilerdeki herhangi bir hatanın düzeltilmesini isteme hakkında da bulunmaktadır. Eğer bu konularda bir isteğiniz olursa doktorunuzla görüşünüz.

Vermiş olduğunuz onaydan vazgeçerseniz, doktorunuz çalışma verilerinizi artık kullanamayacak ya da hiç kimseyle kimliğiniz gizli olsa dahi paylaşamayacaktır.

### ARAŞTIRMA SONUNDA BANA BİLGİ VERİLECEK Mİ?

Talep ettiğinizde değerlendirme sonuçlarınız sözel olarak sizinle paylaşılacak olup, ölçeklerden elde edilecek niceliksel veriler hakkında size geribildirim yapılacaktır.

HER TÜRLÜ SORUNUZLA İLGİLİ İLETİŞİM KURUBİLECEĞİNİZ SORUMLU KİŞİLER:

Dr. Öğr. Üyesi Funda Arun 05327494542

Arş. Gör Dt. Emine Taşkın 05069674172

YENİ BİLGİLER ÇALIŞMADAKİ ROLÜMÜ NASIL ETKİLEYEBİLİR?

Çalışma sürerken ortaya çıkmış olan bütün yeni bilgiler size derhal iletilecektir.

#### GÖNÜLLÜ KATILIM BEYANI

Bu araştırmaya katılma kararımı tamamen gönüllü olarak veriyorum. Bu çalışmaya katılmayı reddedebileceğimi veya katıldıktan sonra istediğim zaman ayrılma hakkımın hiçbir sorumluluk almadan var olduğunu biliyorum. Bu durumun, sağlık kurumunda göreceğim bakım ve tedaviler etkilenmeyeceğinin bilincindeyim. Çalışmadan herhangi bir zamanda ayrılırsam, ayrılma nedenlerimi, ayrılışımın sonuçlarını ve izleyen dönemde alacağım tedavileri doktorumla birlikte değerlendireceğim.

### ÇALIŞMAYA KATILMA ONAYI

Yukarıdaki tüm açıklamaları doktorumla ayrıntılı olarak görüştüm ve kendisi tedavim hakkındaki bütün sorularımı cevapladı. Bu bilgilendirilmiş olur belgesini okudum ve anladım. Bu araştırmaya katılmayı hiçbir baskı altında olmadan kabul ediyor ve bu olur belgesini kendi hür irademle imzalıyorum. Bu onayın, yasal haklarımı koruyan hiçbir mevzuat hükmünü geçersiz kılmadığını biliyorum. Doktorum, saklamam için bu belgenin bir kopyasını ve çalışma sırasında dikkat edeceğim hususları içeren belgeyi bana teslim etmiştir.

| Hastanın Adı Soyadı: | Tarih: | İmza: |
|----------------------|--------|-------|

| Varsa | | |
|----------------------------|--------|-------|
| Veli/Vasinin Adı Soyadı: | Tarih: | İmza: |
| Açıklamaları yapan | | |
| Araştırmacının Adı Soyadı: | Tarih: | |